CLINICAL TRIAL: NCT01320384
Title: Clinical Effect of the Association of Noninvasive Ventilation and High Flow Nasal Oxygen Therapy in Resuscitation of Patients With Acute Lung Injury. A Randomised Study (FLORALI Study)
Brief Title: Clinical Effect of the Association of Noninvasive Ventilation and High Flow Nasal Oxygen Therapy in Resuscitation of Patients With Acute Lung Injury (FLORALI Study)
Acronym: FLORALI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Poitiers university hospital, CHU Poitiers
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FLORALI
Record Dates: First submitted 2010-10-07; First posted 2011-03-22 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Acute Lung Injury; Acute Respiratory Failure
Keywords: ALI
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- O2 conventional : standard low flow therapy (Active Comparator): in order to obtain a SpO2>92%
  Interventions: Other: O2 conventional
- O2-HNF : high flow nasal oxygen therapy (Experimental): set between 30 to 50 l/min,adjusted in order to obtain a SpO2 >92%.
  Interventions: Device: O2-HFN : high flow nasal oxygen therapy
- O2-HFN/NPPV (Experimental): cycling of NIV and O2-HDN
  Interventions: Device: O2-HFN/NPPV : association of high flow nasal oxygen therapy and non invasive positive pressure ventilation

INTERVENTIONS:
Other: O2 conventional — standard low flow therapy
  Arms: O2 conventional : standard low flow therapy
Device: O2-HFN : high flow nasal oxygen therapy — The patient will receive high flow nasal of humidified oxygen, set between 30 to 50 l/min. The inspired fraction of oxygen (FiO2) will be adjusted in order to obtain a SpO2 >92%.
  Arms: O2-HNF : high flow nasal oxygen therapy
Device: O2-HFN/NPPV : association of high flow nasal oxygen therapy and non invasive positive pressure ventilation — The patient will receive successively in a day NPPV and O2-HFN. The NPPV will be applied with an airway humidification achieved by using a heated humidifier and a facial mask adapted to the morphology of the patient. The settings will be adjusted as follow : an inspiratory pressure between 6 to 14 cmH2O, in order to obtain a tidal volume between 7 to 10 ml/kg of predicted weight, a positive expiratory pressure between 0 to 10 cmH2O in order to obtain a SpO2 >92% with the minimal FiO2.
  Arms: O2-HFN/NPPV

SUMMARY:
The aim of the study is to compare, in patients with acute respiratory failure/acute lung injury the efficacy of three different methods of oxygenation to prevent endotracheal intubation :

1. conventional oxygen therapy (O2 conventional)
2. high flow nasal oxygen therapy (O2-HFN)
3. association of high flow nasal oxygen therapy with non invasive positive pressure ventilation (O2-HFN/NPPV).

ELIGIBILITY:
Inclusion Criteria:

* Hypoxemic and no hypercapnic acute respiratory failure :
* severe dyspnea at rest with a respiratory rate >25 breaths/min
* PaO2/FiO2 <300
* PaCO2 <45 mmHg,

Exclusion Criteria:

* age <18 years
* NPPV contraindications
* past history of respiratory chronic disease (COPD, cystic fibrosis…)
* cardiac pulmonary edema
* Pre-defined intubation
* other than respiratory organ failure : systolic pressure <90 mmHg,current treatment with epinephrine or norepinephrine, decreased level of consciousness ( Glasgow score ≤ 12)
* profound aplasia (white cells count <1000/mm 3)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2011-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To compare the number of patients in each group who require endotracheal intubation with mechanical ventilation | at day 28

SECONDARY OUTCOMES:
mechanical ventilation-free to day 28 | 28 days
ICU morbidity | at day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Poitiers University Hospital, Poitiers, France

REFERENCES:
- [Derived] Demoule A, Baptiste A, Thille AW, Similowski T, Ragot S, Prat G, Mercat A, Girault C, Carteaux G, Boulain T, Perbet S, Decavele M, Belin L, Frat JP; from the REVA Network (Research Network in Mechanical Ventilation). Dyspnea is severe and associated with a higher intubation rate in de novo acute hypoxemic respiratory failure. Crit Care. 2024 May 23;28(1):174. doi: 10.1186/s13054-024-04903-5. PMID 38783367
- [Derived] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908